CLINICAL TRIAL: NCT01083979
Title: Intravesical Liposomes for Ulcerative Cystitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kenneth Peters, MD (Other)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-021
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Liposomes; Administration, Intravesical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liposomes (Experimental): Intravesical instillation of Liposomes in sterile water totally 40 cc at four weekly treatments.
  Interventions: Drug: Liposomes

INTERVENTIONS:
Drug: Liposomes — Intravesical instillation
  Other Names: Bladder instillation

SUMMARY:
The objective is to instill liposomes reconstituted with sterile water into the bladder as a compassionate use treatment in one patient with ulcerative interstitial cystitis (IC).

DETAILED DESCRIPTION:
A physician sponsored Investigation New Drug (IN) has been acquired from the FDA for compassionate use of this non-approved treatment in one patient from Dr. Peters' private practice. Since this treatment has not been used previously in the US, we propose to evaluate the safety and efficacy of the treatment in this one patient by comparing pre and post treatment symptom changes.

Prior to treatment (visit 1) baseline measures will be assessed: vital signs,pelvic/bladder pain on a visual analog scale (VAS; "0" being none and "10" being severe), concomitant medications, Serum pregnancy test and Antiphospholipid Antibody Panel, Urine cytology, urinalysis (dipstick), and culture.

At visits 2-5 (4 treatment visits) questionnaires will be completed and vital signs, pain VAS, post void residual (measured by bladder scan or catheter), unanticipated events, and voiding history (voiding diary) will also be assessed. Additionally, cystoscopy will be done prior to the first treatment to view the bladder lining. At each treatment visit, the patients will have a solution of liposomes instilled in the bladder with a catheter, retained for 30 minutes, and be carefully monitored for at least 1 hour after the liposomes are drained.

After treatment, visits 6 and 7 (follow up) will include vital signs with VAS pain assessment, post void residual (PVR), urinalysis (dipstick), unanticipated events assessment, questionnaire completion and review of voiding diary. Visit 8 (study exit) will include the same parameters measured at follow up visits 6 and 7 with the addition of cystoscopy and Antiphospholipid Antibody Panel testing.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative IC for at least 6 months documented,
* Negative urine cytology,
* Able to independently complete self administered questionnaires and voiding diaries.

Exclusion Criteria:

* Pregnant or lactating,
* History of bleeding diathesis,
* On anticoagulant therapy,
* Active peptic ulcer disease,
* Obvious neurological impairment,
* Known allergy to liposomes.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomes
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Liposomes
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Symptom and Problem Severity
Description: The primary objective is to determine the impact of 4 weekly bladder instillations of liposomes on symptoms in one patient with ulcerative interstitial cystitis (IC). The primary endpoint will be assessed at the end of the study, 8 weeks after the last bladder instillation, and will be measured by the O'Leary-Sant IC Symptom and Problem Indices (ICSI-PI) questionnaire. The ICSI is composed of 4 questions that address the occurrence of IC symptoms, specifically urinary urgency, frequency, nocturia, and bladder pain. Scores range from 0 (Not at All) to 5 (Almost Always). The IC Problem Indices questionnaire is also composed of 4 questions. Each question asks the patient to indicate how big a problem each of the 4 symptoms are to them. Scores range from 0 (No Problem) to 4 (Big Problem). Responses to all 8 questions are added together to create a total ICSI-PI score. The total ICSI-PI scores ranges from 0 to 36. A lower score indicates less IC symptoms and/or related problem
Time Frame: Baseline to 12 weeks
Measure: Number; unit: units on a scale
Groups:
- Liposomes: Intravesical instillation of Liposomes in sterile water totalling 40 cc at four weekly treatments.
Arm/Group | Liposomes
Number analyzed (Participants) | 1
units on a scale
  Baseline Total ICSI-PI Score | 22
  12 Week Total ICSI-PI Score | 13

2. Secondary Outcome: Bladder Appearance
Description: The secondary objective to assess treatment efficacy will compare the number of bladder ulcers pre-treatment to the number of ulcers visualized at 12 weeks, the end of the study.
Time Frame: Baseline to 12 Weeks
Measure: Number; unit: Ulcers
Arm/Group | Liposomes
Number analyzed (Participants) | 1
Ulcers
  Total Number of Ulcers at Baseline | 3
  Total Number of Ulcers at 12 Weeks | 0

ADVERSE EVENTS:
Arm/Group | Liposomes
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
This was a single-subject treatment study. Therefore the data analysis and results are limited and are not generalizable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes